CLINICAL TRIAL: NCT06944236
Title: Prevalence of Cardiovascular-Kidney-Metabolic (CKM) Syndrome and Its Relationship With SCORE-2 Risk Score and Body Roundness Index (BRI): A Study From Gaziantep, Turkey
Brief Title: CKM Syndrome Prevalence and Its Association With SCORE-2 and BRI
Acronym: CKM-PREV
Status: Not yet recruiting | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Yildiz Büyükdereli Atadag, Asst. Prof., University of Gaziantep
Other Study IDs: 2025/30
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Syndrome; Cardiovascular Diseases; Chronic Kidney Disease(CKD)
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Renal Insufficiency, Chronic | interventions — Risk Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: All eligible participants aged 30-79 years enrolled from a single family health center in Gaziantep, Türkiye. All participants will undergo anthropometric measurements and be classified into CKM Syndrome stages (0-4) based on clinical and laboratory data. This is a single-group observational study; subgrouping will occur only during analysis.
  Interventions: Other: No intervention is applied. This is a non-interventional, observational study. Anthropometric measurements and existing laboratory data are used for CKM staging and risk assessment.

INTERVENTIONS:
Other: No intervention is applied. This is a non-interventional, observational study. Anthropometric measurements and existing laboratory data are used for CKM staging and risk assessment. — No intervention is applied. This is a non-interventional, observational study. Anthropometric measurements and existing laboratory data are used for CKM staging and risk assessment.

SUMMARY:
This cross-sectional study aims to determine the prevalence of Cardiovascular-Kidney-Metabolic (CKM) syndrome in a community-based adult population in Gaziantep, Türkiye. In addition to estimating the prevalence across CKM stages, the study investigates the associations between CKM syndrome and two key risk indicators: the SCORE-2 cardiovascular risk score and Body Roundness Index (BRI). Findings from this study will provide valuable insights into early cardiometabolic risk profiling and support the development of regionally tailored prevention strategies.

DETAILED DESCRIPTION:
Cardiovascular diseases, diabetes, and chronic kidney diseases are among the leading causes of morbidity and mortality both globally and in Türkiye [1]. The Cardiovascular-Kidney-Metabolic (CKM) Syndrome, which defines the shared pathophysiological basis of these conditions, was classified in 2023 by the American Heart Association (AHA) using a stage-based system ranging from 0 to 4 [1,2]. This study aims to present, for the first time from Türkiye, community-based prevalence data on CKM Syndrome within the framework of this new definition.

In a large-scale cross-sectional study conducted in the United States by Zhu et al. in 2024 [3], CKM stages were found to be associated with social determinants such as education, income, housing, and employment. However, to date, no field study has been conducted in Türkiye based on the AHA's CKM staging system.

This study will also examine the correlation between CKM stages and both the SCORE-2 risk score and the Body Roundness Index (BRI). SCORE-2, developed by the European Society of Cardiology, is a reliable model for estimating 10-year cardiovascular risk based on age, sex, smoking status, systolic blood pressure, total cholesterol, and HDL levels [4,5]. BRI is a novel anthropometric parameter that more sensitively reflects abdominal obesity than body mass index (BMI) [6,7].

With these objectives, the study will:

Provide the first community-based field data on CKM stages in Türkiye,

Reveal the relationships between CKM stages, SCORE-2, and BRI,

Generate locally relevant findings to inform primary care practices.

By demonstrating the usability of test data already obtained within the scope of the Disease Management Platform (HYP), the study will offer a cost-effective model.

In conclusion, this study will provide pioneering data for both the epidemiological assessment and practical management of CKM syndrome screening in Türkiye.

CKM Staging (Stage 0-4) is defined as follows [2]:

Stage 0 - Low Risk Individuals with no identifiable risk factors; considered healthy.

Stage 1 - Early Risk

Presence of at least one metabolic risk factor:

Overweight or obesity (particularly abdominal obesity)

Prediabetes (elevated fasting glucose or HbA1c)

Poor dietary habits and low physical activity

Elevated-normal blood pressure (prehypertension)

Low HDL and/or high triglycerides

Stage 2 - High Risk / Subclinical Disease Individuals with multiple metabolic risk factors but without clinically diagnosed cardiovascular or kidney disease.

Typical combinations in this stage may include:

Dyslipidemia + Prediabetes + Abdominal obesity

Stage 3 - Established Disease

Individuals with a diagnosis of one or more of the following:

Type 2 diabetes

Hypertension

Chronic kidney disease (eGFR < 60 mL/min/1.73 m²) But who have not yet experienced a major cardiovascular event

Stage 4 - Cardiovascular Outcome

Individuals diagnosed with atherosclerotic cardiovascular disease (ASCVD), including:

Myocardial infarction

Stroke

Peripheral artery disease

Basic Data Required for CKM Staging:

Anthropometric Measurements:

Body Mass Index (BMI), waist circumference, neck circumference, waist-to-height ratio, Body Roundness Index (BRI)

Biochemical Tests:

Fasting glucose, HbA1c, lipid profile (HDL, LDL, total cholesterol, triglycerides), creatinine, estimated glomerular filtration rate (eGFR)

Clinical History:

Presence or absence of diagnosed diabetes, hypertension, or chronic kidney disease

History of major cardiovascular events

Methods Study Design and Setting This is a descriptive, community-based field study to be conducted among individuals registered at the Bağlarbaşı Family Health Center, located in the Şahinbey district of Gaziantep, Türkiye. The primary aim of the study is to determine the prevalence of Cardiovascular-Kidney-Metabolic (CKM) Syndrome stages (Stage 0 to 4) among individuals aged 30 to 79 years, and to evaluate the association of these stages with SCORE-2 risk scores and anthropometric indicators.

Study Duration and Site The study will be conducted over a period of six months and will take place at a single site: Bağlarbaşı Family Health Center.

Population and Sample Size The target population includes individuals aged 30 to 79 years who are registered with the Bağlarbaşı Family Health Center. Only individuals with available biochemical test results (including fasting glucose, HbA1c, lipid profile, creatinine, eGFR, and albumin/creatinine ratio) obtained within the last month as part of routine care and accessible via the Disease Management Platform (HYP) will be included.

The total registered population of the center is approximately 35,000 individuals. Based on previous studies reporting a CKM prevalence of approximately 25%, and considering known population size, a minimum sample size of 262 participants was calculated using a 95% confidence level and 5% margin of error. However, to allow meaningful analysis across all five CKM stages, the target sample size has been increased to at least 400 individuals.

Data Collection Only age and sex information will be collected directly from participants. Biochemical data will be accessed via the HYP system. Anthropometric measurements will be obtained on-site by trained healthcare staff.

Anthropometric Measurements

The following measurements will be performed:

Height (cm): Measured using a stadiometer, without shoes, in an upright position.

Weight (kg): Measured using a digital scale, with participants wearing light clothing and no shoes.

Waist Circumference (cm): Measured using a tape measure at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest (spina iliaca anterior superior).

Neck Circumference (cm): Measured at the level of the larynx.

In addition to direct measurements, the following indices will be calculated:

Body Mass Index (BMI) = kg / m²

Waist-to-Height Ratio = waist circumference / height

Body Roundness Index (BRI): Calculated using waist circumference and height, BRI reflects visceral adiposity. It will be computed using a digital Excel-based calculator.

Formula: Based on WC (waist circumference) and H (height)

Biochemical Parameters

Biochemical test results performed within the last month and available via the Disease Management Platform (HYP) will include:

Fasting glucose (mg/dL)

HbA1c (%)

Total cholesterol, LDL, HDL, triglycerides (mg/dL)

Creatinine (mg/dL)

eGFR (mL/min/1.73 m²)

Urine albumin-to-creatinine ratio (if available)

CKM Staging Participants will be classified according to the Cardiovascular-Kidney-Metabolic (CKM) staging algorithm (Stage 0-4) proposed by the American Heart Association (AHA, 2023). Staging will be based on clinical diagnoses and laboratory values obtained within the past month.

CKM Stages Defined:

Stage 0: Healthy individuals with no obesity, metabolic abnormalities, or kidney disease.

Stage 1: Individuals with increased waist circumference and/or BMI ≥ 25 kg/m², along with early metabolic abnormalities such as prediabetes.

Stage 2: Individuals diagnosed with metabolic conditions such as type 2 diabetes, hypertension, or dyslipidemia and/or moderate kidney disease (e.g., eGFR 30-59 mL/min/1.73 m² or presence of proteinuria).

Stage 3: Individuals with high-risk chronic kidney disease (e.g., eGFR <30) or subclinical but high-risk cardiovascular conditions.

Stage 4: Individuals with established clinical cardiovascular disease, such as coronary artery disease, myocardial infarction, stroke, or heart failure.

SCORE-2 Risk Calculation The SCORE-2 algorithm, recommended by the European Society of Cardiology (ESC), will be used to calculate the 10-year cardiovascular risk. It incorporates age, sex, systolic blood pressure, smoking status, total cholesterol, and HDL cholesterol.

As Türkiye is classified as a high-risk region, the following tool will be used:

https://heartscore.escardio.org/Calculate/quickcalculator.aspx?model=high

Note: SCORE-2 is not a fixed formula that can be calculated manually by all users.

It is based on Cox regression models, includes coefficients that vary by sex and country risk level, and must be calculated using the ESC's online calculator or SCORE-2 risk charts.

Key Parameters Used in SCORE-2 Calculation:

Age (30-69 years: SCORE-2; 70-89 years: SCORE-2 OP)

Sex (Female / Male)

Systolic Blood Pressure (mmHg)

Smoking Status (Yes / No)

Total Cholesterol (mg/dL or mmol/L)

HDL Cholesterol (mg/dL or mmol/L)

LDL Cholesterol (mg/dL or mmol/L)

Data Sources for Staging and Risk Assessment All diagnostic and laboratory parameters used in the CKM staging process will be retrieved from participants' existing medical records and test results available through the Disease Management Platform (HYP).

HYP is a national digital health platform designed to facilitate early detection of chronic diseases at the secondary prevention level and guide evidence-based screening and diagnosis for healthcare professionals.

Outcome Measures Both the SCORE-2 cardiovascular risk score and the Body Roundness Index (BRI) will be calculated. These measures will be evaluated as variables associated with CKM staging. Correlation and predictive value analyses will be conducted to assess their relationship with CKM stages.

Inclusion Criteria:

Aged between 30 and 79 years

Having completed the following laboratory tests within the past month:

Fasting glucose

HbA1c

Lipid profile (total cholesterol, LDL, HDL, triglycerides)

Creatinine

Estimated glomerular filtration rate (eGFR)

Residing in Gaziantep, Türkiye

Providing informed consent

Exclusion Criteria:

Individuals with severe physical or mental disabilities

Hospitalization due to an acute illness within the past 3 months

Pregnancy

ELIGIBILITY:
Inclusion Criteria Age between 30 and 79 years Residence in Gaziantep, Türkiye

Availability of the following laboratory tests performed within the past 1 month:

Fasting glucose HbA1c Lipid profile (total cholesterol, LDL, HDL, triglycerides) Creatinine Estimated glomerular filtration rate (eGFR) Ability to provide informed consent

Exclusion Criteria Presence of severe physical or mental disability Hospitalization due to acute illness within the past 3 months Pregnancy

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study will include individuals aged 30 to 79 years who are registered at Bağlarbaşı Family Health Center, located in the Şahinbey district of Gaziantep, Türkiye. The study population represents a community-based sample receiving routine primary care services. Participants will be selected based on the availability of recent laboratory test results (within the past month) from the national Disease Management Platform (HYP). Anthropometric measurements will be obtained on-site. The population reflects a typical adult primary care population in an urban setting.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of CKM Syndrome stages (0-4) | At the time of enrollment (single visit)
  The proportion of participants classified into CKM Syndrome stages 0 to 4 based on AHA 2023 criteria, using clinical, biochemical, and anthropometric data.

SECONDARY OUTCOMES:
Association between CKM stages and SCORE-2 risk scores, BRI | At the time of enrollment (single visit)
  Correlation analysis between CKM stages and BRI values derived from waist circumference and height. Evaluation of the relationship between CKM stage and 10-year cardiovascular risk estimated by SCORE-2 calculator, using ESC criteria for high-risk countries.

CONTACTS AND LOCATIONS:
Locations (1):
- Bağlarbaşı Family Health Center, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the observational nature of the study and the absence of an established data sharing infrastructure.

REFERENCES:
- [Background] Kiremitli T, Kiremitli S, Ulug P, Dinc K, Uzel K, Arslan YK. Are the body shape index, the body roundness index and waist-to-hip ratio better than BMI to predict recurrent pregnancy loss? Reprod Med Biol. 2021 May 21;20(3):327-333. doi: 10.1002/rmb2.12388. eCollection 2021 Jul. PMID 34262401
- [Background] Zhang X, Ma N, Lin Q, Chen K, Zheng F, Wu J, Dong X, Niu W. Body Roundness Index and All-Cause Mortality Among US Adults. JAMA Netw Open. 2024 Jun 3;7(6):e2415051. doi: 10.1001/jamanetworkopen.2024.15051. PMID 38837158
- [Background] Karakayali M, Pusuroglu H, Altunova M, Yilmaz E, Gullu A. Predictive Value of the SCORE, SCORE2, and Pooled Cohort Risk Equation Systems in Patients with Hypertension. Turk Kardiyol Dern Ars. 2023 Sep;51(6):407-414. doi: 10.5543/tkda.2023.74249. PMID 37671521
- [Background] SCORE2 working group and ESC Cardiovascular risk collaboration. SCORE2 risk prediction algorithms: new models to estimate 10-year risk of cardiovascular disease in Europe. Eur Heart J. 2021 Jul 1;42(25):2439-2454. doi: 10.1093/eurheartj/ehab309. PMID 34120177
- [Background] Zhu R, Wang R, He J, Wang L, Chen H, Niu X, Sun Y, Guan Y, Gong Y, Zhang L, An P, Li K, Ren F, Xu W, Guo J. Prevalence of Cardiovascular-Kidney-Metabolic Syndrome Stages by Social Determinants of Health. JAMA Netw Open. 2024 Nov 4;7(11):e2445309. doi: 10.1001/jamanetworkopen.2024.45309. PMID 39556396
- [Background] Ndumele CE, Rangaswami J, Chow SL, Neeland IJ, Tuttle KR, Khan SS, Coresh J, Mathew RO, Baker-Smith CM, Carnethon MR, Despres JP, Ho JE, Joseph JJ, Kernan WN, Khera A, Kosiborod MN, Lekavich CL, Lewis EF, Lo KB, Ozkan B, Palaniappan LP, Patel SS, Pencina MJ, Powell-Wiley TM, Sperling LS, Virani SS, Wright JT, Rajgopal Singh R, Elkind MSV; American Heart Association. Cardiovascular-Kidney-Metabolic Health: A Presidential Advisory From the American Heart Association. Circulation. 2023 Nov 14;148(20):1606-1635. doi: 10.1161/CIR.0000000000001184. Epub 2023 Oct 9. Erratum In: Circulation. 2024 Mar 26;149(13):e1023. doi: 10.1161/CIR.0000000000001241. PMID 37807924
- [Background] Sebastian SA, Padda I, Johal G. Cardiovascular-Kidney-Metabolic (CKM) syndrome: A state-of-the-art review. Curr Probl Cardiol. 2024 Feb;49(2):102344. doi: 10.1016/j.cpcardiol.2023.102344. Epub 2023 Dec 14. PMID 38103820
- See also: AHA — https://www.heart.org/en/professional/cardiovascular-kidney-metabolic-health